CLINICAL TRIAL: NCT04938505
Title: Assessment of Health Related Quality of Life in Women Who Underwent Breast Reconstruction After Radical Surgery (RMQOL)
Brief Title: Assessment of Health Related Quality of Life in Women Who Underwent Breast Reconstruction After Radical Surgery
Acronym: RMQOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A011828-47
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nowadays, breast reconstruction is an integral care after mastectomy in breast cancer patient.

With the personalized care, choice a breast reconstructive is an important step involving decisions and mutual accord between patients and their physicians in order to anticipate clinical and psychosocial results.

Two main families of breast reconstruction techniques are often performed including advantages and complications impacting health related quality of life.

Routine assessment of health related quality of life in patients underwent breast reconstruction could allow to identify factors of satisfaction o be taken into account in the choice of breast reconstruction technique in order to improve practices and quality of life of patients

ELIGIBILITY:
Inclusion Criteria:

* Normal Breast Checkup ( Mammography, echography and breast magnetic resonance imaging)in the previous 6 months
* French speaking and writing fluency
* Agree to participate after receive all information

Exclusion Criteria:

* Patients with an inability to complete HRQOL questionnaires (cognitive disorders, language barrier)
* Patient with a failed first breast reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing breast reconstruction after mastectomy for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-04 (Actual); Primary Completion 2024-05-04 (Estimated); Study Completion 2025-05-04 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life scores assessed by Breast Q questionnaire | 12 months after breast reconstruction

SECONDARY OUTCOMES:
Number of anxious and depress participants as assessed by Hospital Anxiety and Depression Scale (HADS) | 12 months after breast reconstruction
  HADS has 14 items rated from 0 to 3 and covers 2 dimensions. Seven questions related to the anxiety dimension and seven other related to the depressive dimension, yielding 2 scores, A (Anxiety) and D (Depression). The maximum score for each dimension is 21. A score of 11 or higher indicates the probable presence of the disorder.
social support as assessed by Sarason's Social Support Questionnaire 6-item (SSQ6) | 12 months after breast reconstruction
  Social support is measured across 2 dimensions: support availability, through the number of contacts that the patient can count on (0 to 9 people) and quality of support, through patient satisfaction with support received. Each item represents a situation in which the patient may need support. Patient is asked to cite the number of people that she could count on in that particular situation. Concerning the second item, the patient is asked to assess satisfaction with the support provided. The scores are generated according to Sarason's recommendations. A score is calculated for each dimension. Support availability score is calculated as the sum of the number of people available for the 6 items, this score ranges from 0 to 54, with 54 representing the highest availability. The social support satisfaction score is calculated by the sum of the satisfaction of the 6 items. This score ranges from 6 to 36, with 36 representing the highest level of satisfaction
level of the precariousness and the disparities of health at breast reconstruction patient by the questionnaire Evaluation of the Precariousness and the Disparities of Health for the Centers of Examination of Health (EPICES) | 12 months after breast reconstruction
  EPICES is used to assess individual level of the precariousness. It includes 11 items and generate precariousness score from 0 to 100. Patient which a score EPICES >30 is considered as having a high level of precariousness
Health related quality of life scores assessed by Breast Q questionnaire | 24 months after breast reconstruction
Health related quality of life scores assessed by Breast Q questionnaire | 36 months after breast reconstruction
Health related quality of life scores assessed by Breast Q questionnaire | 48 months after breast reconstruction
Health related quality of life scores assessed by Breast Q questionnaire | 60 months after breast reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Clementine JANKOWSKI, MD, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- Centre Georges Francois Leclerc, Dijon, France